CLINICAL TRIAL: NCT04120038
Title: Self-Management for Amputee Rehabilitation Using Technology (SMART) Phase 2
Brief Title: Self-Management for Amputee Rehabilitation Using Technology
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other); GF Strong Rehabilitation Centre (Other)
Responsible Party: Principal Investigator, William C. Miller, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H19-02241
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Unilateral Trans Tibial/Femoral Lower Limb Amputation
Keywords: Occupational Therapy; Rehabilitation; Lower-Limb Amputations; Amputees; Telehealth; Remote Rehabilitation; Telerehabilitation; E-learning; Education; Self-Management; Ambulation; Coping Strategies; Outcomes; Prevalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART & Peer Support (Experimental)
  Interventions: Device: Self-Management for Amputee Rehabilitation using Technology [SMART]

INTERVENTIONS:
Device: Self-Management for Amputee Rehabilitation using Technology [SMART] — Participants will complete a 6-week tablet-based education program for individuals with LLA that will provide them with self-management education.

SUMMARY:
The purpose of this study is to determine the effect of 6 weeks of the SMART Program on the walking capacity and confidence of individuals with unilateral lower limb amputation (LLA). Our primary hypothesis is that SMART can improve walking capacity in individuals with LLA. Our secondary hypothesis is that SMART can improve ambulation confidence, body function, depression, body image, pain, balance confidence, activities of daily living, satisfaction with life and habit formation for skin monitoring and prosthetic cleaning in individuals with LLA. A post-intervention one on one interview will be conducted to understand SMART acceptability. The entirety of the study, including intervention administration, assessment, and interviews will be conducted online.

DETAILED DESCRIPTION:
Participants will receive an online link to access the SMART platform. Online training on using the SMART platform will be provided for participants. Participants will be asked to complete one education module per week at their own convenience and weekly online meetings with a peer over the 6-week intervention period. The educational modules include psychological adaptation, residual limb management, nutrition/weight control, managing a prosthetic limb, managing chronic conditions and enhancing mobility. The modules include instructional movies, goal setting logs, and quizzes. A module can be stopped or "re-wound" at any point, and the participant's place and work-to-date is automatically saved. The SMART platform will be asynchronously monitored through a web portal by the trainer, who will be a PhD candidate in Rehabilitation Sciences and observe participant progress and provide feedback if required. If there is no online activity within a 7-day (consecutive) period, the trainer will contact the participant to inquire the reasons for inactivity and troubleshoot any problems including technical issues. Clinical outcomes measures will be collected at two timepoints (T1 & T2). A post-intervention one on one interview will be conducted to explore SMART acceptability.

ELIGIBILITY:
Inclusion Criteria:

1. adults who are 19 years of age or older.
2. individuals who are post unilateral transtibial/transfemoral amputation and casted an initial prosthesis within the past year.
3. English speaking.
4. living in British Columbia or Ontario, Canada.
5. have access to an internet connectable device (e.g., computer or tablet)

Exclusion Criteria:

1) people who are unable to use SMART program (e.g., visual, auditory, cognitive, or physical impairments)

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Timed Up & Go Test (TUG) | 6 weeks
  Functional assessment of walking capacity measured in seconds over 3 meters walkway

SECONDARY OUTCOMES:
Ambulatory Self-Confidence Questionnaire (ASCQ) | 6 weeks
  22-item questionnaire where participants are asked to rate questions on a scale from 0 (not confident at all) to 10( extremely confident)
The Center for Epidemiologic Studies Depression Scale (CES-D) | 6 weeks
  Self-rating measure assessing depression, with final scores ranging from 0 to 60, with total score above 23 indicating clinical depression

OTHER OUTCOMES:
Revised Amputee Body Image Scale (ABIS-R) | 6 weeks
  14-item measure that evaluates self perception of body image in individuals with LLA, exploring their feelings about physical appearance, levels of anxiety and comfort in various social situations after amputation. Total ABIS-R score ranges from 20-100, greater score indicates higher body image disturbance.
Pain Questionnaire | 6 weeks
  A questionnaire will be used to assess both pain frequency and intensity over one week in three categories: residual limb pain (pain in the above portion of the amputated site), phantom limb pain (pain in the missing portion of the limb), and the nonpainful phantom limb sensation (sensations in the missing portion of the limb which were not painful)
Activities Specific Balance Confidence Scale (ABC). | 6 weeks
  16-item self-report measure that assesses perceived balance confidence, which is important for mobility. Total ABC score ranges from 0-100, with greater score indicating higher levels of balance confidence.
Barthel Index (BI) | 6 weeks
  10-item scale that measures independence in self-care and mobility
Satisfaction With Life Scale (SWLS) | 6 weeks
  5-item measure scored on a Likert scale from 1 (strongly disagree) to 7 (strongly agree).
Self-Report Habit Index (SRHI). | 6 weeks
  12-item questionnaire based on the 7-point Likert scale with the range of total score between 0 to 84, which higher scores show the stronger habit strength
Short Musculoskeletal Function Assessment (SMFA) | 6 weeks
  Items 1-34 of an assessment of difficulties with daily activities and experiencing problems because of injury.
Physical Activity Identity (PAI) | 6 weeks
  9-item questionnaire used to assess the extent physical activity is integrated within the concept of self.
Patient Education Material Assessment Tool (PEMAT) | 6 weeks
  26-item questionnaire used to assess the understandability and actionability of an educational intervention from the perspective of participants.
Perceived Usefulness Questionnaire (PUQ) | 6 weeks
  17-item questionnaire used to assess the perceived usefulness, ease-of-use, intention to continue usage, and satisfaction of SMART.

CONTACTS AND LOCATIONS:
Overall Officials: William C Miller, PhD, Principal Investigator — University of British Columbia
Locations (1):
- GF Strong Rehabilitation Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273